CLINICAL TRIAL: NCT03767998
Title: The Manifestation of Surface EMG of Swallowing Muscles in Stroke Patients With Respiratory Muscle Training. A Prospective Study.
Brief Title: The Manifestation of Surface EMG of Swallowing Muscles in Stroke Patients With Respiratory Muscle Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMRPG8F0961
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Cerebrovascular Disorders
Keywords: Respiratory muscle training; Spirometry; Maximal Inspiratory Pressure; Maximal Expiratory pressure; Surface electromyography
MeSH Terms: conditions — Cerebrovascular Disorders | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IMST group (Experimental): Interventions: Respiratory muscle training for IMST. Inspiratory muscle training for patients with inspiratory muscle weakness (MIP less than 70% of normal range). IMT will commence from 30% to 60 % of MIP and then adjust one level of training loading according to the tolerance of continuously breathing through a respiratory trainer for two sets of 30 breaths or 6 sets of 10 repetitions with one or two minute of rest between sets, once per day, 5 days per week.
  Interventions: Other: Respiratory muscle training for IMST; Other: Regular Rehabilitation
- Control group (Active Comparator): Intervention: Non-training group, receive regular rehabilitation. All participants will receive usual rehabilitation care including body positioning instruction, postural correction, breathing control, cough maneuver, respiratory muscle stretch, chest wall mobility exercise and ventilation, fatigue management.
  Interventions: Other: Regular Rehabilitation
- EMST group (Experimental): Intervention: Respiratory muscle training for EMST. For patients with only swallowing disturbance. Training resistance will be adjusted accordingly. The loading will be performed with the previous resistance setting or even lower if training load is not tolerated or not completed.
  Interventions: Other: Regular Rehabilitation; Other: Respiratory muscle training for EMST

INTERVENTIONS:
Other: Respiratory muscle training for IMST — 2 sets of 30 breaths or 6 sets of 10 repetitions with one or two minute of rest between sets, once per day, 5 days per week, training with breathing trainer.
  Arms: IMST group
Other: Regular Rehabilitation — Regular Rehabilitation: 2-3 times a week, 6 weeks.
Other: Respiratory muscle training for EMST — 5 sets, 5 repetition with one or two minute of rest between sets, twice per day, 5 days per week, training with breathing trainer.
  Arms: EMST group

SUMMARY:
Purpose: To investigate of the respiratory function and swallowing function after respiratory muscle training, and the manifestation of surface EMG of swallowing muscles, and the lateralization of placement of electrodes in stroke patients. Methods: A prospective study. Consecutive patients with diagnosis of stroke will be proved by magnetic resonance image or computerized tomography. Stroke patients, aged 35-80 years old, with inspiratory muscle weakness or swallowing disturbance will be enrolled and randomly divided into control group (usual rehabilitation alone) and experimental group (inspiratory muscle strengthening training (IMST) group for patients with inspiratory muscle weakness and expiratory muscle strengthening training (EMST) for patients with swallowing disturbance, respectively. Each patients will receive usual rehabilitation. In the meanwhile we will recruit 23 healthy subjects for the control group.

Each patient will receive baseline characteristics, duration of stroke, Brunnstrom's stage, muscle power, spirometry, peak cough flow, maximal inspiratory pressure (MIP),maximal expiratory pressure (MEP), resting heart rate, perception of dyspnea, resting oxyhemoglobin saturation (SpO2), hand grip strength of unaffected upper limb. And patients with swallowing disturbance will receive swallowing screen test, Functional Oral Intake Scale to evaluate the functional level of oral intake of food and liquid, and voice quality analysis for voice quality and bilateral surface electromyography for measurement of masseter, oris orbicularis, submental muscle and infraspinatus muscles. All of patients will be assessed again at 6 weeks and 12 weeks later.

Patient with respiratory muscle weakness will receive IMT from 30% to 60 % of MIP through a respiratory trainer for two sets of 30 breaths or 6 sets of 10 repetitions. For patients with swallowing disturbance, EMST will commence from 15% to 75% of threshold load of an individual's MEP, 5 sets, 5 repetition with one minute of rest between sets.. The training resistance will be adjusted accordingly, with one or two minute of rest between sets. Both group will receive respiratory training, twice per day, 5 days per week. For checking the compliance of RMT at home, patients will be monitored by making a phone call to them once a week.

DETAILED DESCRIPTION:
Stroke patients commonly to have respiratory muscle weakness and swallowing disturbance. Their cardiorespiratory function could be markedly impaired within 7 weeks after a stroke, and maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) reduced. Dysphagic patients usually had reduced hyolaryngeal excursion. The contraction of submandibular hyolaryngeal muscles (geniohyoid, mylohyoid, anterior digastric) and thyohyoid muscles can influence on the hyoid bone and largynx . The decreased excursion and elevation of hyolaryngeal complex has been considered as one of cause of penetration and aspiration in patients with dysphagia.

Respiratory muscle training (RMT) could improve cough effectiveness and reduce the incidence of pneumonia in acute stroke. RMT could significantly increase in MIP and MEP with training intensity of inspiratory muscle training (IMT) varied from 30% to 60% of MIP, duration of 3 to 7 times per week and duration of each session from 10-30 minutes for a period of training from 6 to12 weeks in subacute stroke patients.

Expiratory muscle strength training (EMST) had potential benefit for respiratory muscle strength, swallowing and cough function. EMST could significantly increase duration of activation with higher peak amplitudes of EMG signal of the submental muscles as compared to dry and wet swallowing in stroke patients(Wheeler, et al. 2007) and it also had promising outcomes for airway protection in persons with dysphagia second to neuromuscular impairment.

Swallowing phase including oral phase, pharyngeal phase, pharyngeal and initial esophageal pahased. Surface EMG (sEMG), a simple, noninvasive, radiation-free and reliable method, can be used to screen and differentiate the swallowing disturbance by recording activity of surface EMG over the swallowing muscles, including orbicularis oris, masseters, submental muscles and infrahyoid muscles. The electric activity of sEMG can be filtered and rectified as EkG-looking line. It can provide complementary information to assess the dysphagia.

Correlation of sEMG signals during swallowing in healthy adults has been reported And stroke patients with middle cerebral artery infarction had delayed swallowing onset, pretrigger duration of hyoid bone. The sEMG showed shorter duration of sEMG activity, latency between the start of EMG activity and actual movement, shortened submental muscle activity, and prolonged pretrigger duration during swallowing.

Hypothesis Respiratory muscle training can activate the respiratory muscles, stimulate motor cortex of central nervous system of speech, swallowing and respiratory function through the certain process of neuroplasticity in brain and spinal cord. EMST could facilitate submental muscle contraction, increase submental muscle force and elevate the hyolaryngeal complex during swallowing.

However, rare reports regarding the relationship between the respiratory muscle training and swallowing dysfunction in stroke patients. And stroke patients with different lesions may have specific sEMG patterns; the differentiation of sEMG pattern of swallowing muscles in different stroke disease with dysphagia is not explored yet, and also short of standards to study the sEMG of swallowing muscles.

In this study, we will use a simple respiratory muscle training device(Threshold type) to train respiratory muscles and follow up its effect on swallowing, cough, voice quality in stroke patients with respiratory muscle weakness and/or swallowing disturbance.

Forty-six stroke patients with respiratory muscle weakness, age between 35 to 80 years, will be enrolled. The participants will be randomly assigned by a computer random number generator into two groups, including the experimental group (RMT group plus usual rehabilitation) and the control group (usual rehabilitation alone). All allocations will be concealed in the opaque envelopes. The research assistant will enroll the participants, generate the allocation sequence, and assign participants to their groups after obtaining the informed consent.

The patient will be randomized into 3 groups:

Group I: IMST only: inspiratory muscle training for patients with inspiratory muscle weakness (MIP less than 70% of normal range).

Group II: EMST: for patients with swallowing disturbance.

Group III: Control group will receive regular rehabilitation.

Each subject with respiratory muscle weakness or swallowing disturbance, baseline characteristics, including height, weight, body mass index, duration of the disease, neurological level (Brunnstrom's stage), spirometry, peak cough flow, resting heart rate, systolic and diastolic blood pressure, resting oxyhemoglobin saturation (SpO2), MIP, MEP, Borg's scale (0.5 to 10), 6-minute walking test, cough function, fatigue assessment scale and caregiver stress scale. Pulmonary function and respiratory muscle strength will be assessed by an experienced technician in our pulmonary functional room as a baseline at the begin of training program, and at end of program(6 weeks).

Training protocol:

Group I: IMST only:

IMT will commence from 30% to 60 % of MIP and then adjust one level of training loading according to the tolerance of continuously breathing through a respiratory trainer for two sets of 30 breaths or 6 sets of 10 repetitions with one or two minute of rest between sets, once per day, 5 days per week. Training resistance will be adjusted as tolerated. The loading will be performed with the previous resistance setting or even lower if training load is not tolerated or not completed.

During IMT, patients will be instructed to place their lips around breathing trainer in a sitting position with a nose-clip, inhale with enough force to open the valve (inhale deeply and forcefully), exhale through the mouthpiece (exhale slowly and gently), and then continue inhaling and exhaling without removing the device from their mouths. The training load and training program will be instructed by an experienced respiratory technician.

Group II: EMST: for patients with only swallowing disturbance EMST will commence from 15% to 75% of threshold load of an individual's MEP, 5 sets, 5 repetition with one or two minute of rest between sets, twice per day, 5 days per week. And training resistance will be adjusted accordingly. The loading will be performed with the previous resistance setting or even lower if training load is not tolerated or not completed. Each patients with swallowing disturbance will receive swallowing screen test, Functional Oral Intake Scale, voice quality analysis and surface electromyography by an experience physician and experienced speech therapist to evaluate the functional level of oral intake of food and liquid, voice quality and measurement of submental muscle strength respectively. And swallowing training program will be conducted by an experienced speech therapist.

GroupIII：Control group will receive regular rehabilitation.

Outcome measurements:

Each subject's baseline characteristics, including height, weight, body mass index, and duration of the disease, neurological level (Brunnstrom's stage), spirometry, resting heart rate, rest respiratory rate, blood pressure, resting oxyhemoglobin saturation (SpO2), MIP, MEP, or the lowest resting SpO2, Borg's scale, six-minute walk work value and distance, six-minute upper extremity ergometry, peak cough flow, non-affected upper limb strength, fatigue assessment scale etc.

For rectified and filtered sEMG, swallowing duration (the time lapse between the start and the end of swallowing. In second), mean peak amplitude (inμsec), and shape of contraction patterns of different stage of swallowing will be analyzed.

The timing of serial evaluation including the assessment at baseline, 6 weeks and 3 month later.

ELIGIBILITY:
Inclusion Criteria:

* Patients identified as stroke,
* Diagnosed by magnetic resonance image or computerized tomography
* Capable of performing voluntary respiratory maneuvers

Exclusion Criteria:

* Increased intracranial pressure
* Uncontrolled hypertension
* Complicated arrhythmia
* Decompensated heart failure
* Unstable angina
* Myocardial infarction in the preceding 3 months
* Pneumothorax
* Bullae/blebs
* Severe cognitive function
* Emotional disturbance
* Infection

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
MIP (maximal inspiratory pressure) | At the beginning and the end of program respectively, up to 6 weeks.
  MIP(cm H20) is measured after maximal expiration while patients sitting and wearing a nose-clip. For MIP, more negative pressure is better.
MEP (maximal expiratory pressure) | At the beginning and the end of program respectively, up to 6 weeks.
  MEP(cm H20) is measured after maximal inspiration while patients sitting and wearing a nose-clip. For MEP, more positive is better.
Surface EMG data | At the beginning and the end of program respectively, up to 6 weeks.
  The EMG of masseter, orbicularis oris, submental (anterior belly of digastrics, mylohyoid, geniohyoid) and infrahyoid muscles will be recorded. Three trials of dry swallowing, voluntary water swallowing, and breathing through a breathing trainer in low intensity and about 50% of the measured intensity of maximal expiratory pressure at beginning of program will be recorded

SECONDARY OUTCOMES:
Forced vital capacity, FVC(liter) | At the beginning and the end of program respectively, up to 6 weeks.
  Pulmonary functional test, the determination of the vital capacity from a maximally forced expiratory effort.
Forced vital capacity, FVC(%pred)(liter) | At the beginning and the end of program respectively, up to 6 weeks.
  Pulmonary functional test, the determination of the vital capacity from a maximally forced expiratory effort.
Forced expiratory volume 1/Forced vital capacity, FEV1/FVC(%) | At the beginning and the end of program respectively, up to 6 weeks.
  Pulmonary functional test, a calculated ratio used in the diagnosis of obstructive and restrictive lung disease.
Maximal mid-expiratory flow, MMEF(%) | At the beginning and the end of program respectively, up to 6 weeks.
  Pulmonary functional test, the peak of expiratory flow as taken from the flow-volume curve and measured in liters per second.
Peak cough flow(liter/min) | At the beginning and the end of program respectively, up to 6 weeks.
  Maximum speed of expiration.
Resting heart rate | At the beginning and the end of program respectively, up to 6 weeks.
  Heart rate of patient during resting.
Resting respiratory rate | At the beginning and the end of program respectively, up to 6 weeks.
  Respiratory rate of patient during resting.
Functional Oral Intake Scale | At the beginning and the end of program respectively, up to 6 weeks.
  Level 1: Nothing by mouth. Level 2: Tube dependent with minimal attempts of food or liquid. Level 3: Tube dependent with consistent oral intake of food or liquid. Level 4: Total oral diet of a single consistency. Level 5: Total oral diet with multiple consistencies, but requiring special preparation or compensations.Level 6: Total oral diet with multiple consistencies without special preparation, but with specific food limitations. Level 7: Total oral diet with no restrictions. Level 1 to level 7.
Borg's Scale | At the beginning and the end of program respectively, up to 6 weeks.
  Modified Borg scale (0.5 to 10) 0 Nothing at all 0.5 Very, very slight (just noticeable)
  1. Very slight
  2. Slight
  3. Moderate
  4. Somewhat severe
  5. Severe
  7 Very severe 8 9 Very, very severe (almost maximal) 10 Maximal
Fatigue Assessment Scale | At the beginning and the end of program respectively, up to 6 weeks.
  Score: 5-50. 1 = Never, 2 = Sometimes; 3 = Regularly; 4 = Often and 5 = Always. 10 items.

CONTACTS AND LOCATIONS:
Overall Officials: Liaw Mei-Yun, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation, Kaohsiung Chang Gung Memorial Hospital., Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No